CLINICAL TRIAL: NCT00077402
Title: A Phase 2 Study Of Fenretinide In Patients With Hormone Refractory Prostate Cancer
Brief Title: Fenretinide In Treating Patients With Advanced or Metastatic Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Therapeutics Research Group (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CTRG-P18/02; CDR0000350305 (Registry Identifier: PDQ (Physician Data Query)); NCI-6062
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2006-12

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fenretinide

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well fenretinide works in treating patients with advanced or metastatic hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of fenretinide, in terms of the prostate-specific antigen (PSA) response rate, in patients with advanced or metastatic hormone-refractory prostate cancer.

Secondary

* Determine the objective response rate in patients with identifiable soft tissue disease treated with this drug.
* Determine the duration of PSA response in patients treated with this drug.
* Determine PSA progression-free survival of patients treated with this drug.
* Determine overall survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine self-rated symptoms, functions, attitudes to oral therapy, and quality of life of patients treated with this drug.

OUTLINE: This is a multicenter, open-label study.

Patients receive oral fenretinide twice daily on days 1-7. Treatment repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each course, and at the end of therapy.

PROJECTED ACCRUAL: Approximately 21-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Measurable or non-measurable disease
  * Metastatic disease allowed
* Castrate levels of serum testosterone (either after orchiectomy or maintained on a luteinizing hormone-releasing hormone agonist or antagonist)
* Prostate-specific antigen (PSA) greater than 10 ng/mL at baseline and rising, with 2 consecutive increases measured at least 1 week apart*
* No known brain metastases NOTE: *If the third PSA value has not risen above the second PSA value, a fourth measurement must be obtained that is higher than the second value

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* AST and ALT no greater than 2.5 times upper limit of normal
* Bilirubin normal

Renal

* Creatinine normal OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Able to tolerate oral medication
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to fenretinide
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 6 weeks since prior antiandrogen therapy with any of the following:

  * Cyproterone
  * Flutamide
  * Bicalutamide
  * Nilutamide
* Concurrent corticosteroids allowed provided therapy was initiated before study entry

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy, including for pain
* No concurrent radioisotopes (e.g., strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium)

Other

* More than 4 weeks since prior investigational agents
* No concurrent antioxidants (e.g., ascorbic acid or vitamin E), vitamin A, or beta carotene supplements
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial anticancer agents or therapies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Response rate as measured by RECIST at ≥ 9 weeks

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTC

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boyer, Study Chair — Sydney Cancer Centre at Royal Prince Alfred Hospital
Locations (6):
- Australia (2):
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Singapore (3):
  - Cancer Institute at National University Hospital, Singapore
  - National Cancer Centre - Singapore, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore

REFERENCES:
- [Result] Moore MM, Stockler M, Lim R, Mok TS, Millward M, Boyer MJ. A phase II study of fenretinide in patients with hormone refractory prostate cancer: a trial of the Cancer Therapeutics Research Group. Cancer Chemother Pharmacol. 2010 Oct;66(5):845-50. doi: 10.1007/s00280-009-1228-x. Epub 2010 Jan 16. PMID 20082080